CLINICAL TRIAL: NCT01643642
Title: A Efficacy and Cost-effectiveness Study of a Brief Interventions for Mood and Anxiety Disorders: Brief Intake, Treatment and Routine Outcome Monitoring (ROM)
Brief Title: Cost- Effectiveness Study of Brief Interventions for Mood and Anxiety Disorders
Acronym: K&K
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: GGZ Rivierduinen (Other)
Responsible Party: Principal Investigator, D. Meuldijk, PhD Student, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P09.146/NL29380.058.09; P09.146/NL29380.058.09 (Other: CME LUMC/Toetsingonline ABR-formulier)
Record Dates: First submitted 2011-09-08; First posted 2012-07-18 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Depressive Disorder; Anxiety Disorder
MeSH Terms: conditions — Depressive Disorder; Anxiety Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive behavioral treatment/farmacotherapy intervention (Experimental): Brief intervention; intake, cognitive behavioral treatment/farmacotherapy (SSRI) and ROM
  Interventions: Other: Cognitive behavioral treatment/farmacotherapy intervention
- Treatment As Usual (Other): Control group, TAU
  Interventions: Other: Treatment As Usual

INTERVENTIONS:
Other: Cognitive behavioral treatment/farmacotherapy intervention — Brief cognitive behavioral intervention/farmacotherapy; intake, treatment and ROM
  Arms: Cognitive behavioral treatment/farmacotherapy intervention
Other: Treatment As Usual — Other: Treatment As Usual
  Arms: Treatment As Usual

SUMMARY:
This study compares both clinical effectiveness and cost-effectiveness of a brief, intensified therapy and diagnostic method for patients with mood and/or anxiety disorders with Treatment As Usual (TAU) at five outpatient Mental Healthcare Centers in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* Male of female adolescents
* Adolescents aged between 18 to 65 year
* Adolescents main complaint: Mild to moderate anxiety and/or mood disorders with or without psychiatric and/or somatic co-morbidity
* Adolescents with proper understanding of the Dutch language.

Exclusion Criteria:

* Adolescents with current psychotic or bipolar traits,
* Adolescents with homicidal or suicidal risk
* Adolescents with severe social disfunctioning
* No proper understanding of the Dutch language

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the intervention | approximately 3 years (start: march 2010).
  Effectiveness of the intervention is investigated by the main questionnaires: Web Screening Questionnaire (WSQ) and Brief Symptom Inventory (BSI) as conducted by ROM

SECONDARY OUTCOMES:
Cost-effectiveness intervention | approximately 3 years (start: march 2010).
  Cost-effectiveness is explored by an open questionnaire Trimbos/iMTA Questionnaire for Cost Associated with Psychiatric Illness (TIC-P).
  Additionally patient and therapist satisfaction about the intervention is explored.

CONTACTS AND LOCATIONS:
Locations (1):
- Rivierduinen, South Holland, Netherlands

REFERENCES:
- [Derived] Meuldijk D, Carlier IV, van Vliet IM, van Veen T, Wolterbeek R, van Hemert AM, Zitman FG. The clinical effectiveness of concise cognitive behavioral therapy with or without pharmacotherapy for depressive and anxiety disorders; a pragmatic randomized controlled equivalence trial in clinical practice. Contemp Clin Trials. 2016 Mar;47:131-8. doi: 10.1016/j.cct.2015.12.021. Epub 2016 Jan 5. PMID 26762883